CLINICAL TRIAL: NCT03012217
Title: Prospective Clinical Evaluation of the FilmArray Respiratory Panel 2 (RP2)
Brief Title: Prospective Clinical Evaluation of the FilmArray Respiratory Panel 2
Acronym: RP2
Status: Completed | Type: Observational
Sponsor: BioFire Diagnostics, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: DX-SDY-026541
Record Dates: First submitted 2017-01-03; First posted 2017-01-06 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Upper Resp Tract Infection
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasopharyngeal swabs.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Specimens that meet inclusion criteria
  Interventions: Other: Observational Study

INTERVENTIONS:
Other: Observational Study

SUMMARY:
This is a performance study to test the sensitivity and specificity of the BioFire FilmArray Respiratory Panel (RP) 2. The purpose of this study is to prospectively collect and test residual NPS specimens and generate performance data to support regulatory classification of the FilmArray RP2 as an in vitro diagnostic (IVD) in the US, European Union (EU), Canada, and other regions.

DETAILED DESCRIPTION:
The FilmArray Respiratory Panel 2 (RP2) is an automated sample-to-answer PCR-based diagnostic for the identification of common upper respiratory viral and bacterial pathogens in nasopharyngeal swab (NPS) specimens collected in viral transport media (VTM). The purpose of this study is to prospectively collect and test residual NPS specimens and generate performance data to support regulatory classification of the FilmArray RP2 as an in vitro diagnostic (IVD) in the US, European Union (EU), Canada, and other regions.

Clinical performance evaluations will be initiated at sites in the US and/or EU during the 2016/2017 respiratory illness season, approximately September through December.Prior to performing the prospective clinical evaluation, each participating site will have the necessary Institutional Review Board (IRB) reviews (or equivalent for non-U.S. sites).

Specimens for inclusion in this study will be residual, de-identified NPS collected in VTM leftover from clinician-ordered respiratory pathogen testing.

Comparator testing will be performed using de-identified specimen aliquots at a central reference laboratory.

This study is funded by BioFire Diagnostics, LLC. The FilmArray device conforms to the requirements of the European Union In Vitro Diagnostic Directive (IVDD). This study was designed such that every precaution has been taken to protect the health and safety of patients, users, and other persons.

ELIGIBILITY:
Inclusion Criteria:

* Specimen is residual NPS in VTM left over from standard of care testing under clinician order for respiratory pathogen analysis
* Specimen has been held at appropriate temperature
* Sufficient volume remaining after standard of care testing and available for use in the study

Exclusion criteria:

* Specimen other than NPS in VTM (e.g. nasopharyngeal aspirate, anterior or midturbinate swab, oropharyngeal swab, NPS collected in medium other than VTM)
* Specimen cannot be tested within the defined storage parameters
* Insufficient specimen volume for testing

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Only residual NPS specimens from patients with clinician-ordered respiratory pathogen testing will be enrolled.
Sampling Method: Probability Sample
Enrollment: 1612 (Actual)
Dates: Start 2016-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
sensitivity and specificity of device | 3 months

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Loyola University Medical Center, Maywood, Illinois
  - Nationwide Children's Hospital, Columbus, Ohio
  - Primary Children's Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No